CLINICAL TRIAL: NCT05016687
Title: A Randomised, Double-blind, Single-centre, Placebo-controlled, First-in-human Clinical Trial Evaluating the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of CUR-N399 in Healthy Volunteers.
Brief Title: First-in-human Clinical Trial Evaluating CUR-N399 in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curovir AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CURCT-001
Record Dates: First submitted 2021-07-02; First posted 2021-08-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Enterovirus Infections; Rhinovirus
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Enterovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental Part I Cohort 1-5: CUR-N399 (Experimental): Healthy subjects 18-55 years will receive single ascending doses of CUR-N399. Planned doses for respective Cohorts: Cohort 1: 2.5 mg, Cohort 2: 7.5 mg, Cohort 3: 17.5 mg, Cohort 4: 35 mg, Cohort 5: 50 mg.
  Interventions: Drug: CUR-N399
- Experimental Part I Cohort 1-5: Placebo (Placebo Comparator): Healthy subjects will receive Placebo to match treatment of CUR-N399.
  Interventions: Drug: Placebo
- Experimental Part IIa Cohort 1-3: CUR-N399 (Experimental): Healthy subjects 18-55 years will receive multiple ascending doses of CUR-N399 during a 7-day period. Planned doses for respective Cohorts: Cohort 1: 10 mg/day, Cohort 2: 25 mg/day, Cohort 3: 50 mg/day.
  Interventions: Drug: CUR-N399
- Experimental Part IIa Cohort 1-3: Placebo (Placebo Comparator): Healthy subjects 18-55 years will receive Placebo to match CUR-N399 treatment during a 7-day period.
  Interventions: Drug: Placebo
- Experimental Part IIb: CUR-N399 (Experimental): Healthy subjects >/= 65 years will receive multiple ascending doses of CUR-N399 during a 7-day period. The dose to be administered will determined based on safety results in Part IIa.
  Interventions: Drug: CUR-N399
- Experimental Part IIb: Placebo (Placebo Comparator): Healthy subjects >/= 65 years will receive Placebo to match CUR-N399 treatment during a 7-day period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CUR-N399 — CUR-N399 will be administered as oral capsules.
  Arms: Experimental Part I Cohort 1-5: CUR-N399; Experimental Part IIa Cohort 1-3: CUR-N399; Experimental Part IIb: CUR-N399
Drug: Placebo — Placebo capsules matching CUR-N399 will administered.
  Arms: Experimental Part I Cohort 1-5: Placebo; Experimental Part IIa Cohort 1-3: Placebo; Experimental Part IIb: Placebo

SUMMARY:
The purpose of the trial is to evaluate CUR-N399, a PI4KB inhibitor, in a first-in-human trial to evaluate the safety, tolerability and pharmacokinetics profile of single and multiple ascending doses in healthy adults.

In the SAD part of the trial, single oral doses of CUR-N399 will be administered in 5 sequential cohorts. In all cohorts, safety and PK will be assessed before and after dose. Exploratory nasopharyngeal swab for assessment of airway infectants will be performed before dose and in the morning of Day 3.

In SAD part Cohort 4: A urine sample will be taken from the first morning void on Day 1 and urine will be collected for potential quantification of CUR-N399 (and metabolites) during the first 24 hours post-dose.

The MAD part of the trial will explore multiple ascending dosing of CUR-N399. The initial dose, dose escalation and dosing schedule will be based on emerging knowledge of safety, tolerability and PK of CUR-N399 observed in the SAD part of the trial. CUR-N399 will be administered in 3 sequential cohorts. An additional MAD cohort will evaluate CUR-N399 in older adults ≥65 years.

All SAD and MAD cohorts will evaluate 8 subjects. Within each cohort, subjects will be randomised in a 3:1 ratio to receive CUR-N399 (n=6) or placebo (n=2) in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Part I and IIa: Healthy male or female subject aged 18-50 years inclusive. Part IIb: Healthy male or female subject aged ≥65 years inclusive.
3. Body Mass Index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2.
4. Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
5. WOCBP must practice abstinence (only allowed when this is the preferred and usual lifestyle of the subject) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 4 weeks after last dose. Female subjects must refrain from donating eggs from the date of dosing until 3 months after dosing with the IMP. Their male partner must agree to use a condom during the same time frame if he has not undergone vasectomy.

Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] 25-140 IE/L is confirmatory).

Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP. Their female partner of child-bearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above). -

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
3. Current or history of gastrointestinal bleedings, inflammatory bowel disease, irritable bowel syndrome or coeliac disease, as judged by the Investigator.
4. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
5. Any planned major surgery within the duration of the study.
6. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and HIV.
7. After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges: Part I, IIa: Systolic blood pressure <90 or >140 mmHg, or Diastolic blood pressure <50 or >90 mmHg, or Pulse <40 or >90 beats per minute (bpm) Part IIb: Systolic blood pressure <90 or >160 mmHg, or Diastolic blood pressure <50 or >100 mmHg, or Pulse <40 or >90 bpm
8. Prolonged QTcF (>450 ms for men, >470 ms for women), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
9. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to CUR-N399.
10. Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within 2 weeks prior to the (first) administration of IMP, at the discretion of the Investigator. NB. The use of a stable dose of levothyroxine is allowed for subjects in Part IIb.
11. Any use of omeprazole products (or products of the same drug class) within 2 weeks prior to the (first) administration of IMP, at the discretion of the Investigator.
12. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Subjects consented and screened but not dosed in previous Phase I studies are not excluded.
13. Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
14. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to (first) administration of the IMP.
15. History or presence of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
16. Presence or history of drug abuse, as judged by the Investigator.
17. History of, or current use of, anabolic steroids.
18. Excessive caffeine consumption defined by a daily intake of >5 cups of caffeine containing beverages.
19. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
20. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
All Parts: Adverse events (AE) | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Incidence (frequency, intensity and seriousness) of AEs
All Parts: Clinically significant changes in electrocardiograms (ECGs) | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Single 12-lead ECG will be recorded in supine position after 10 minutes of rest using an ECG machine. HR and PR, QRS, QT and QTcF intervals will be recorded.
All Parts: Clinically significant changes in vital signs (pulse) | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Pulse will be recorded.
All Parts: Clinically significant changes in vital signs (blood pressure) | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Blood pressure will be recorded.
All Parts: Clinically significant changes in safety laboratory parameters (clinical chemistry) | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Blood samples for analysis of clinical chemistry parameters:
  * Alanine aminotransferase (ALT)
  * Albumin
  * Alkaline phosphatase (ALP)
  * Aspartate aminotransferase (AST)
  * Bilirubin (total and conjugated)
  * Calcium
  * Cholesterol (HDL, LDL, total)
  * Creatinine (estimated Glomerular Filtration Rate [eGFR] included)
  * C-reactive protein (CRP)
  * Glucose
  * Lactate dehydrogenase (LD)
  * Phosphate
  * Potassium
  * Sodium
  * Triglycerides
  * Urea
  will be collected and sent to the certified clinical chemistry laboratory and analysed by routine analytical methods.
All Parts: Clinically significant changes in safety laboratory parameters (heamatology) | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Blood samples for analysis of haematology parameters:
  * Haematocrit
  * Haemoglobin (Hb)
  * Platelet count
  * Red blood cell (RBC) count
  * White blood cell (WBC) count with differential count
  will be collected and sent to the certified clinical chemistry laboratory and analysed by routine analytical methods.
All Parts: Clinically significant changes in safety laboratory parameters (coagulation) | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Blood samples for analysis of coagulation parameters:
  * Activated Partial Thromboplastin Time (APTT)
  * Prothrombin Complex International Normalised Ratio (PK[INR])
  will be collected and sent to the certified clinical chemistry laboratory and analysed by routine analytical methods.
All Parts: Clinically significant changes in physical examinations | From start of treatment Day 1 to End of Study (Day 8 SAD and Day 14 MAD)
  • Routine physical examinations will be performed. Incidence of clinically significant changes will be recorded.

SECONDARY OUTCOMES:
All Parts: Pharmacokinetics (PK) of CUR-N399 (AUC0-t) | Pre-dose Day 1 to 48 hours post last dose (Day 3 SAD and Day 9 MAD respectively)
  Area under the curve (AUC) from time 0 to time t (AUC0-t)
All Parts: Pharmacokinetics (PK) of CUR-N399 (AUC0-∞) | Pre-dose Day 1 to 48 hours post last dose (Day 3 SAD and Day 9 MAD respectively)
  AUC from time 0 to infinity (AUC0-∞)
All Parts: Pharmacokinetics (PK) of CUR-N399 (T½) | Pre-dose Day 1 to 48 hours post last dose (Day 3 SAD and Day 9 MAD respectively)
  Terminal half-life (T½)
All Parts: Pharmacokinetics (PK) of CUR-N399 (Cmax) | Pre-dose Day 1 to 48 hours post last dose (Day 3 SAD and Day 9 MAD respectively)
  Observed maximum plasma concentration (Cmax)
All Parts: Pharmacokinetics (PK) of CUR-N399 (Tmax) | Pre-dose Day 1 to 48 hours post last dose (Day 3 SAD and Day 9 MAD respectively)
  Time to Cmax (Tmax)
All Parts: Pharmacokinetics (PK) of CUR-N399 (dose proportionality) | Pre-dose Day 1 to 48 hours post last dose (Day 3 SAD and Day 9 MAD respectively)
  Dose proportionality (based on AUC and Cmax)
All Parts: Pharmacokinetics (PK) of CUR-N399 (CL/F) | Pre-dose Day 1 to 48 hours post last dose (Day 3 SAD and Day 9 MAD respectively)
  Apparent total body clearance following extravascular administration (CL/F)
All Parts: Pharmacokinetics (PK) of CUR-N399 (Vz/F) | Pre-dose Day 1 to 48 post last dose (Day 3 SAD and Day 9 MAD respectively)
  Apparent volume of distribution following extravascular administration (Vz/F)
Part II a+b: Pharmacokinetics (PK) of CUR-N399 (AUCtau) for MAD groups | After first dose (Day 1) and up to 48 hours post last dose (Day 9)
  AUC for the dosing interval (AUCtau)
Part II a+b: Pharmacokinetics (PK) of CUR-N399 (Ctrough) for MAD groups | Pre-dose administration on Days 2 to 7
  Observed concentration at the end of a dosing interval (Ctrough)
Part II a+b: Pharmacokinetics (PK) of CUR-N399 (Accumulation ratio) for MAD groups | Day 1 to 48 hours post last dose (Day 9)
  Accumulation ratio

OTHER OUTCOMES:
All parts: Nasopharyngeal swabs to evaluate airway infectants | Pre-dose Day -1 to Day 3
  Nasopharyngeal swab samples will be taken to evaluate the presence and levels of a panel of airway infectants:
  * Respiratory syncytial virus
  * Metapneumovirus
  * Influenza a, b
  * All 4 Coronaviruses
  * Adenovirus
  * Parainfluenza virus 1, 2, 3
  * Mycoplasma
  * Clostridium difficile
  * Pneumococci
Part I Cohort 4: CUR-N399 (and metabolites) in urine in SAD Cohort | Pre-dose Day 1 to Day 3
  Potential quantification of unchanged CUR-N399 and metabolites in urine
Part II a+b: Metabolic profile of CUR-N399 in plasma in MAD groups | Day 1 to Day 9
  Potential future metabolite identification in plasma and possible comparison with metabolite exposure in pre-clinical safety studies (metabolites in safety testing [MIST])
Part II a+b: To assess age-related differences in safety of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | From Start of Treatment Day 1 to End of Study Day 14
  To assess age related incidence (frequency and severity) of AEs
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (AUC0-t) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Pre-dose to 48 hours after first dose (Day 3) and after last dose Day 7 to 48 hours post-dose (Day 9)y 1 to 24 hours post last dose Day 8
  To assess age related differences in AUC0-t
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (AUCtau) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Pre-dose Day 1 to 48 hours post last dose Day 9
  AUC for the dosing interval (AUCtau)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (T½) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | After first dose Day 1 and up to 48 hours after last dose Day 9
  Terminal half-life (T½)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (Tmax) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Up to 48 hours after first dose Day 1 (Day 3) and last dose Day 7 (Day 9)
  Time to Cmax (Tmax)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (Cmax) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Up to 48 hours after first dose Day 1 (Day 3) and last dose Day 7 (Day 9)
  Observed maximum plasma concentration (Cmax)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (Dose proportionality) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Up to 48 hours after first dose Day 1 (Day 3) and last dose Day 7 (Day 9)
  Dose proportionality (based on AUCtau and Cmax)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (Ctrough) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Pre-dose of last dose Day 7
  Observed concentration at the end of a dosing interval (Ctrough)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (CL/F) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Up to 48 hours post last dose Day 7 (Day 9)
  Apparent total body clearance following extravascular administration (CL/F)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (Vz/F) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Up to 48 hours post last dose Day 7 (Day 9)
  Apparent volume of distribution following extravascular administration (Vz/F)
Part II a+b: To assess age-related differences in pharmacokinetic (PK) profile (Accumulation ratio) of two age groups 18-55 vs ≥65 year in MAD Cohort with Older adults | Up to 48 hours post last dose Day 7 (Day 9)
  Accumulation ratio

CONTACTS AND LOCATIONS:
Overall Officials: Nina Lindblom, PhD, Study Director — Curovir AB
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden